CLINICAL TRIAL: NCT06634966
Title: Segmentectomy for Solid-dominant GGO-featured Invasive Lung Cancer With Size of 2-3cm: a Single-arm, Multi-center, Phase III Trial
Brief Title: Segmentectomy for Solid-dominant Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Haiquan Chen, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1025
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Segmentectomy; Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Segmentectomy (Experimental): Segmentectomy is performed for solid-dominant invasive lung cancer with size of 2-3cm.
  Interventions: Procedure: Segmentectomy

INTERVENTIONS:
Procedure: Segmentectomy — The lungs are divided into multiple lobes. A segmentectomy involves the removal of part of one of the lobes of the lung to entirely remove a cancerous tumor. segmentectomy can preserve more normal functional lung tissues.
  Other Names: Segment resection

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1025. The goal of this clinical trial is to confirm the theraputic effect of segmentectomy for solid-dominant invasive lung cancer with size of 2-3cm. The main questions it aims to answer are:

* The 5-year disease-free survival of patients having solid-dominant invasive lung cancer with size of 2-3cm;
* The post-operative lung function tests after receiving segmentectomy. Participants will receive segmentectomy as the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent form and are willing to complete the study according to the plan;
* Aged from 18 to 80 years old;
* ECOG equals 0 or 1;
* Not receiving lung cancer surgery before;
* Confirmed to be invasive lung adenocarcinoma intraoperatively or postoperatively;
* Ground glass-dominant lung nodules
* Consolidation-to-tumor ratio (CTR) ranges from 0.5 to 1, and tumor size ranges from 2 to 3cm;
* cN0 without distant metastasis;
* Tumors could be completely resected assed by surgeons;
* Not receiving chemotherapy or radiotherapy before.

Exclusion Criteria:

* CTR is not 0.5-1, or size is not 2-3cm;
* Tumors could not be completely resected assed by surgeons;
* Not lung adenocarcinoma diagnosed cytologically or pathologically;
* Receiving lung cancer surgery before;
* Receiving radiotherapy or chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival | 5 years
  The event is defined as the tumor recurrence or the death due to any causes.

SECONDARY OUTCOMES:
Lung function test | Half year and one year after surgical resection
  FEV1/FVC ratio
5-year overall survival | 5 years
  The event is defined as death due to any causes or last follow-up.
The site of tumor recurrence and metastasis | From date of surgery to the last follow-up or date of death from any cause, whichever came first, assessed up to 5 years.
  Outpatient follow-up was conducted regularly after surgery, and the recurrence or metastasis site and time will be recorded.
Segmentectomy completion rate | From the beginning of the surgery to the end of the surgery.
  Proportion of patients who complete planned segmentectomy.
Radical segmentectomy (R0 resection) completion rate | From surgery to the release of the final pathology report, an average of two weeks.
  According to the postoperative pathology report of the patients, the proportion of patients with no residual tumor after radical segmentectomy accounted for all patients who underwent segmentectomy.
Surgery-related complications | From surgery to patient discharge or 30 days after surgery.
  such as air leak, atrial fibrillation, intraoperative or postoperative hemorrhage, postoperative infection, bronchopleural fistula, etc

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China